CLINICAL TRIAL: NCT07180134
Title: Effects of Health Informatics for Symptom Management and Resistance Exercise Strategies on Quality of Life and Sarcopenia in Post-Esophagectomy Patients With Esophageal Cancer: A Mixed-Methods Study
Brief Title: Health Informatics and Resistance Exercise for Symptom Management and Quality of Life in Post-Esophagectomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Ling Chang, Assistant Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202302087B0
Record Dates: First submitted 2025-08-19; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Cancer (EsC); Sarcopenia; Quality of Life
Keywords: Esophagectomy; Nutrition; Quality of life; Exercise
MeSH Terms: conditions — Esophageal Neoplasms; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: the experimental group also received a 12-week intervention consisting of "symptom management health informatics" and "home-based resistance exercise with elastic bands." The health informatics component included educational videos and an instant communication platform addressing common postoperative gastrointestinal symptoms, their mechanisms, and management strategies, such as reflux, dysphagia, dumping syndrome, and delayed gastric emptying. The communication platform enabled two-way interaction, allowing patients to raise concerns and health providers to respond promptly. The resistance exercise program included instructional videos and individualized exercise prescriptions taught before discharge. Patients were instructed to perform band-based resistance exercises at home, avoiding practice within one hour after meals. Each session lasted 40-60 minutes, including warm-up, resistance, and cool-down, performed three times per week for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Participants receive standard postoperative nursing care and education as routinely provided by the clinical team. No additional interventions will be given.
  Interventions: Behavioral: Usual Care Group
- Symptom Management Health Informatics plus Resistance Exercise Group (Experimental): Participants receive access to a symptom management health informatics program and a structured resistance band exercise training program.
  Interventions: Behavioral: symptom management health informatics plus Resistance band exercise training

INTERVENTIONS:
Behavioral: symptom management health informatics plus Resistance band exercise training — Access to educational videos and an instant messaging platform for real-time communication, delivered over 12 weeks.
  plus Structured resistance band exercise, 3 times per week, ~30 minutes per session, for 12 weeks under research team guidance.
  Arms: Symptom Management Health Informatics plus Resistance Exercise Group
Behavioral: Usual Care Group — Standard postoperative nursing care and education routinely provided by the clinical team. No additional interventions will be given.
  Arms: Usual Care Group

SUMMARY:
Participants are invited to take part in a research study. In accordance with the requirements of the health authorities, participants must be informed of the purpose of the study and its potential risks. Participation is voluntary, and each participant is free to decide whether or not to enroll. The study may be discussed with trusted individuals, and sufficient time may be taken to consider the decision. If any part of this consent form is unclear, questions may be directed to the principal investigator or the research team, who will provide an explanation.

If a participant chooses not to participate, appropriate treatment will still be provided. Even if a participant agrees to participate initially, withdrawal is allowed at any time without affecting medical rights or the care that should be received.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with esophageal cancer and having undergone esophagectomy
* Postoperative pathological report confirms R0 resection (complete tumor removal)
* Able to be discharged after surgery
* With or without adjuvant chemoradiotherapy
* Clear consciousness and able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

* Presence of severe cardiovascular disease or psychiatric disorders
* Inability to communicate in Mandarin Chinese or Taiwanese
* Disease progression during the intervention period that prevents continuation of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-C30 score) | Baseline, 1 month, 3 months, 6 months after intervention
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) is a validated and widely used instrument for assessing quality of life in patients with cancer. It includes five functional scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health status/quality of life scale, and several single-item symptom measures (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Scores are linearly transformed to a 0-100 scale; higher scores on functional and global health scales indicate better functioning/quality of life, whereas higher scores on symptom scales indicate greater symptom burden.

SECONDARY OUTCOMES:
Esophageal Cancer-related Symptoms (EORTC QLQ-OES18 score) | 1 month, 3 months, 6 months after intervention
  The EORTC QLQ-OES18 is a validated disease-specific module designed to assess esophageal cancer-related symptoms and treatment side effects. It includes 18 items covering dysphagia, eating restrictions, reflux, pain, trouble swallowing saliva, choking when swallowing, dry mouth, taste problems, cough, and speech difficulties. Each item is scored on a 4-point Likert scale and linearly transformed to a 0-100 scale, with higher scores indicating greater symptom burden.
Sarcopenia Status (e.g., SARC-F or handgrip strength, muscle mass index) | Baseline, 1 month, 3 months, 6 months after intervention
  Sarcopenia risk will be assessed using the SARC-F questionnaire, which evaluates strength, assistance with walking, rising from a chair, climbing stairs, and falls. Each item is scored 0-2, with a total score ranging from 0 to 10. A score ≥4 indicates risk of sarcopenia.
Body Mass Index (BMI) | Baseline, 1 month, 3 months, 6 months after intervention
  Body mass index (BMI) will be calculated as weight in kilograms divided by height in meters squared (kg/m²). Weight will be measured using a calibrated digital scale, and height will be measured with a stadiometer at baseline. Changes in BMI will be assessed at follow-up visits. Lower BMI values after surgery may indicate postoperative weight loss or malnutrition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang YL, Tsai YF, Chao YK, Wu MY. Quality-of-life measures as predictors of post-esophagectomy survival of patients with esophageal cancer. Qual Life Res. 2016 Feb;25(2):465-475. doi: 10.1007/s11136-015-1094-4. Epub 2015 Aug 4. PMID 26238649
- [Background] Chang YL, Tsai YF, Wu YC, Hsieh MJ. Factors relating to quality of life after esophagectomy for cancer patients in Taiwan. Cancer Nurs. 2014 Jan-Feb;37(1):4-13. doi: 10.1097/NCC.0b013e318277dc53. PMID 23357884
- [Background] Chang YL, Tsai YF, Hsu CL, Chao YK, Hsu CC, Lin KC. The effectiveness of a nurse-led exercise and health education informatics program on exercise capacity and quality of life among cancer survivors after esophagectomy: A randomized controlled trial. Int J Nurs Stud. 2020 Jan;101:103418. doi: 10.1016/j.ijnurstu.2019.103418. Epub 2019 Sep 11. PMID 31670173
- See also: Chang Gung University — https://www.cgu.edu.tw/